CLINICAL TRIAL: NCT01432717
Title: A Phase 1 Randomized, Double-Blind, Placebo-Controlled, Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamic Effects of ACE-536 in Healthy Postmenopausal Women
Brief Title: Study of ACE-536 in Healthy Postmenopausal Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Acceleron Pharma, Inc., a wholly-owned subsidiary of Merck & Co., Inc., Rahway, NJ USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A536-02
Record Dates: First submitted 2011-09-01; First posted 2011-09-13 (Estimated); Last update posted 2012-11-07 (Estimated); Status verified 2012-11

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — luspatercept

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ACE-536 (Experimental): Subjects assigned to 1 of 5 possible dosing groups.
  Interventions: Biological: ACE-536
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: ACE-536 — Subjects receive a total of 2 subcutaneous doses of ACE-536 on Day 1 and Day 15.
  Arms: ACE-536
Other: Placebo — Subjects receive a total of 2 subcutaneous doses of placebo on Day 1 and Day 15.
  Arms: Placebo

SUMMARY:
The purpose of this study is to find out whether ACE-536 can be safely given to patients. This study will also look to see if ACE-536 increases red blood cells, the cells that carry oxygen in the body.

ELIGIBILITY:
Key Inclusion Criteria:

* Postmenopausal women
* Body Mass Index (BMI) of 20 - 32 kg/m2.

Key Exclusion Criteria:

* History of hypertension
* Subject has received any erythropoiesis stimulating agents (e.g., Epogen, Procrit, Aranesp, etc.) within 6 months prior to Day 1
* History of clinically significant cardiac, endocrine, hematologic, hepatic, immune, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal, and/or other disease
* Surgery within 3 months (other than minor cosmetic surgery or minor dental procedures)
* Subject has received treatment with another investigational drug, or approved therapy for investigational use within 1 month prior to Day 1, or if the half-life of the previous product is known, within 5 times the half-life prior to Day 1, whichever is longer

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-09; Primary Completion 2012-09 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse Events as a measure of safety and tolerability. | 22 weeks

SECONDARY OUTCOMES:
ACE-536 serum concentration after single and multiple ascending doses. | 22 weeks
Hemoglobin levels after single and multiple ascending doses. | 22 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Acceleron Investigative Site, Tempe, Arizona, United States

REFERENCES:
- [Derived] Attie KM, Allison MJ, McClure T, Boyd IE, Wilson DM, Pearsall AE, Sherman ML. A phase 1 study of ACE-536, a regulator of erythroid differentiation, in healthy volunteers. Am J Hematol. 2014 Jul;89(7):766-70. doi: 10.1002/ajh.23732. Epub 2014 Apr 26. PMID 24715706